CLINICAL TRIAL: NCT06940401
Title: A Phase I/II Clinical Study to Evaluate JS111 Capsules in Patients With Locally Advanced, Metastatic, or Recurrent Non-Small Cell Lung Cancer (NSCLC) Harboring Epidermal Growth Factor Receptor (EGFR) Mutations.
Brief Title: JS111 in Patients With Advanced NSCLC Harboring EGFR Mutations
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suzhou Junjing BioSciences Co., Ltd. (Industry)
Collaborators: Sponsor GmbH (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JS111-003-I/II-NSCLC
Record Dates: First submitted 2025-04-08; First posted 2025-04-23 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-04

CONDITIONS: NSCLC

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- JS111 capsules (AP-L1898) (Experimental): 160 or 240 mg once daily (QD)
  Interventions: Drug: JS111 capsules (AP-L1898)

INTERVENTIONS:
Drug: JS111 capsules (AP-L1898) — In Phase I, approximately 3-12 subjects will be enrolled in each dose group (160 mg QD or 240 mg QD) and receive oral JS111 capsules once daily until any treatment discontinuation criteria are met. After all subjects have completed at least 21 days observation following the first dose, the Safety Monitoring Committee (SMC) will review safety and pharmacokinetic data to make decisions. Phase II will continue enrollment at the RP2D dose level until approximately 30 subjects have been treated at that dose.

SUMMARY:
To evaluate the safety, tolerability, and preliminary efficacy of JS111 capsules in patients with locally advanced, metastatic, or recurrent NSCLC harboring EGFR mutations;to determine the recommended Phase II dose (RP2D).

DETAILED DESCRIPTION:
This is a Phase II clinical study evaluating JS111 capsules (AP-L1898) as monotherapy in patients with advanced NSCLC harboring EGFR mutations.Approximately 3 to 42 treatment-naïve patients with EGFR mutation-positive locally advanced, metastatic, or recurrent NSCLC will be enrolled.Based on prior safety, PK, and efficacy data, two dose levels-160 mg QD and 240 mg QD-will be tested to assess safety, tolerability, PK, and preliminary efficacy, and to determine the recommended Phase II dose (RP2D), as referenced in Section 4.3.

The study includes two parts:

Part 1:

Each dose group will enroll 3-12 subjects who will receive oral JS111 capsules daily until meeting treatment discontinuation criteria. Once all subjects complete at least the Day 21 observation following the first dose 21 days of treatment , the Safety Monitoring Committee (SMC) will review the data to decide whether to:

1. Select RP2D for further enrollment;
2. Continue enrollment for further evaluation;
3. Explore other dose levels;
4. Amend or terminate the study if needed. Subjects who receive <80% of planned doses or discontinue for non-drug-related reasons during the 21-day period will be replaced. Mutation subtypes (exon 19 deletion or exon 21 L858R) will be evenly assigned across dose groups, starting from the lower dose.

Part 2:

Subjects will be enrolled into the RP2D cohort until ~30 patients have been treated with the dose. Subjects from the other group may continue on the same dose or switch to RP2D as appropriate. JS111 will be taken once daily in 21-day cycles to further assess safety, PK, and preliminary efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged ≥18 years at the time of signing informed consent.
2. Histologically or cytologically confirmed locally advanced, metastatic, or recurrent NSCLC that is unresectable and unsuitable for curative chemoradiotherapy.
3. No prior systemic anti-tumor therapy for locally advanced or metastatic NSCLC.
4. Confirmed presence of EGFR-sensitizing mutations (exon 19 deletion or L858R mutation), either alone or co-occurring with other EGFR mutations (including T790M-positive cases). Local laboratory results are acceptable if the test is well-validated, qualified through external quality assessment or molecular diagnostics certification, or approved by NMPA.
5. At least one measurable lesion according to RECIST v1.1.
6. ECOG performance status of 0 or 1.
7. Life expectancy of ≥12 weeks.
8. Adequate function of key organs.
9. Women of childbearing potential (WOCBP) with non-sterilized male partners must have a negative serum pregnancy test within 7 days prior to first dosing and agree to use effective contraception from informed consent signing until 2 months after the last dose.
10. Non-sterilized male subjects with female partners of childbearing potential must agree to use effective contraception (as described in Section 10.3.2) from informed consent signing until 4 months after the last dose and must refrain from sperm donation during this period.
11. Willingness to participate and signed informed consent provided by the subject.

Exclusion Criteria:

1. Presence of any of the following disease conditions.

   a. Histologically or cytologically confirmed small cell lung cancer (SCLC) components, large cell neuroendocrine carcinoma, or sarcomatoid features；b. Conditions that may affect oral drug absorption, distribution, metabolism, or excretion (e.g., inability to swallow, severe vomiting, uncontrolled diarrhea, major GI surgery, Crohn's disease, ulcerative colitis)；c. Known leptomeningeal metastasis；d. Symptomatic brain metastases；e. Uncontrolled pleural effusion, pericardial effusion, or ascites requiring frequent drainage (e.g., ≥ once per month)；f. Untreated or symptomatic spinal cord compression; or previously treated spinal cord compression not stable for at least 4 weeks before enrollment；
2. Prior or concurrent treatments.

   a. Any previous treatment with EGFR-TKIs;b. Use of strong CYP3A inhibitors/inducers within 14 days before the first dose or requirement for such treatment during the study;c. Ongoing treatment with drugs known to prolong QT interval or cause Torsades de Pointes;d. Receipt of any investigational drug within 4 weeks or 5 half-lives (whichever is shorter) before first dosing;e. Concurrent participation in another clinical study, unless it is non-interventional or in follow-up phase;f. Major surgery (e.g., craniotomy, thoracotomy, laparotomy) within 4 weeks before first study drug administration;g. Local radiotherapy within 14 days before the first dose (e.g., palliative radiotherapy for bone metastases);
3. Unresolved toxicities from prior anti-tumor therapy not recovered to ≤ Grade 1 per CTCAE, except for alopecia, Grade 2 peripheral neuropathy, or Grade 2 hypothyroidism judged to be non-risk by the investigator.
4. Known hypersensitivity to study drug or its excipients.
5. Cardiac abnormalities, including.

   a. QTcF ≥450 ms for males or ≥470 ms for females (mean of 3 ECGs during screening);b. Clinically significant arrhythmias (e.g., complete left bundle branch block, 3rd-degree AV block, PR interval >250 ms);c. Risk factors for Torsades de Pointes (e.g., hypokalemia, family history of long QT syndrome or inherited arrhythmias); d. Left ventricular ejection fraction (LVEF) <50%;
6. History or suspected diagnosis of interstitial lung disease, drug-induced pneumonitis, idiopathic pulmonary fibrosis, or other significant pulmonary diseases (except for ≤ Grade 1 radiation pneumonitis).
7. Serious infection (CTCAE > Grade 2) within 4 weeks prior to first dosing, such as pneumonia requiring hospitalization. Active pulmonary inflammation on baseline imaging or infection symptoms requiring antibiotics within 2 weeks prior to dosing (excluding prophylactic use).
8. History of immunodeficiency, including HIV positivity, congenital or acquired immunodeficiency disorders, or history of organ/allogeneic bone marrow transplantation or autologous stem cell transplantation.
9. Active tuberculosis or history of active TB within 1 year prior to enrollment; or untreated TB if diagnosed over 1 year ago.
10. Active hepatitis B (HBsAg positive and HBV DNA ≥500 U/mL) or hepatitis C (anti-HCV positive and HCV RNA above the detection limit).
11. History of other malignancies unless low-risk (5-year survival >90%) and adequately treated, e.g., basal/squamous cell carcinoma of the skin, in situ cervical or breast cancer, localized prostate cancer, or papillary thyroid carcinoma.
12. Pregnant or breastfeeding women, or those planning to become pregnant during the study.
13. Uncontrolled comorbid conditions.
14. Any serious or uncontrolled ocular disease.
15. Any other condition judged by the investigator as potentially leading to early withdrawal from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-04-30 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-11-05 (Estimated)

PRIMARY OUTCOMES:
AE | up to 3years
  Safety endpoints: incidence and severity of adverse events (AE); Abnormal changes in laboratory and other tests with clinical significance
ORR | up to 3years
  ORR
RP2D | up to 3years
  RP2D

SECONDARY OUTCOMES:
PFS | up to 3years
  Progression-free survival (PFS)
DCR | up to 3years
  disease control rate (DCR)
OS | up to 3years
  overall survival (OS)
(Cmax) | up to 6 months
  Evaluation of the first dose peak concentration (Cmax)
(Tmax） | up to 6 months
  Evaluation of the first dose time to peak (Tmax)
(AUC0-t） | up to 6 months
  Evaluation of the area under the concentration-time curve (AUC0-t) for the first dose
(t1/2） | up to 6 months
  Assessment of the first dose elimination half-life (T 1/2)
(CL/F） | up to 6 months
  Assessment of apparent clearance rate of the first dose (CL/F)
(Vd/F） | up to 6 months
  Assessment of apparent volume distribution (Vd/F) for the first dose
(λz） | up to 6 months
  Evaluation of the first dose elimination rate constant (λz)
(Cmin, ss） | up to 6 months
  Assessment of steady-state trough concentration (Cmin, ss) for multiple doses
(Cmax, ss） | up to 6 months
  Assessment of steady-state peak concentration (Cmax, ss) for multiple doses
(Cavg, ss） | up to 6 months
  Assessment of mean steady-state plasma concentrations (Cavg, ss) for multiple doses
Plasma concentrations of JS111 | up to 6 months
  Evaluation of plasma concentrations of JS111
Plasma concentrations of JS111 active metabolite M546b | up to 6 months
  Evaluation of plasma concentrations of JS111 active metabolite M546b

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No